CLINICAL TRIAL: NCT00319982
Title: Treatment of Preclinical Hypertrophic Cardiomyopathy With Diltiazem
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Carolyn Yung Ho, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001936; K23HL078901 (NIH)
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy; Left ventricular hypertrophy; Diltiazem
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular | interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I- Diltiazem (Experimental): Diltiazem- study medication
  Interventions: Drug: Diltiazem
- II- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diltiazem — Sustained release formulation titrated to a target dose of 360 mg daily, or a maximum of 5 mg/kg/day in pediatric subjects for the duration of the study period
  Arms: I- Diltiazem
Drug: Placebo — Placebo comparator (double-blind allocation of study medication)
  Arms: II- Placebo

SUMMARY:
This is a pilot clinical trial to assess whether the administration of diltiazem may be able to decrease the development or progression of hypertrophic cardiomyopathy (HCM). Diltiazem is a commonly used medication for the treatment of high blood pressure and studies on animals with HCM suggest that diltiazem decreases disease development. This study specifically targets individuals in the "prehypertrophic" phase of HCM-- those with documented sarcomere gene mutations without echocardiographic or EKG evidence of LVH, and therefore without a clinical diagnosis of HCM.

The hypothesis of this study is that starting diltiazem administration early in life (in the prehypertrophic phase) will decrease the progression of HCM in individuals with sarcomere gene mutations. This will be assessed by looking at an improvement in the heart's ability to relax using echocardiography, as well as exploratory analyses of a broad range of features reflecting the heart's structure and function.

DETAILED DESCRIPTION:
STUDY RATIONALE:

Hypertrophic cardiomyopathy (HCM) is a genetic disorder characterized by histopathologic findings of cardiac myocyte disarray and fibrosis, and clinical manifestations of unexplained left ventricular hypertrophy (LVH), diastolic dysfunction, and an increased risk for sudden death. It is a common disorder affecting approximately 1 in 1000 individuals in the general population. Dominantly-acting mutations in contractile proteins-genes encoding the elements of the sarcomere apparatus-- have been shown to be the genetic etiology of HCM. Contemporary management strategies for HCM focus on identification of individuals at high risk for sudden death and management of symptoms. There is no current therapy available which address disease prevention or phenotypic attenuation.

Dysregulation of intracellular calcium handling is a fundamental and early manifestation of sarcomere mutations. Animal models of HCM demonstrated abnormal Ca2+ cycling prior to the development of myocyte disarray or hypertrophy. Manipulation of intracellular Ca2+ handling in young, pre-hypertrophic mice with HCM via administration of the L-type Ca2+ channel blocker, diltiazem, attenuated the degree of hypertrophic remodeling and diminished the phenotypic manifestations of sarcomere mutations. Notably, if treatment was initiated later in life, after LVH was allowed to develop, there was no significant effect. Although this strategy has not yet been tested in humans, diltiazem is a commonly-used medication with a long track record of safety and tolerability.

Mutation carriers without discernible echocardiographic left ventricular hypertrophy (designated G+/LVH-) represent a unique population of individuals with early disease who are ideal candidates for preemptive strategies to attempt to attenuate phenotypic development. One clinical marker of early disease is a subtle abnormality of LV diastolic function, detectable by tissue Doppler echocardiography (TDI). Individuals with sarcomere mutations have evidence of abnormal diastolic function by TDI as demonstrated by a 13-19% reduction in early myocardial relaxation velocities (E'), as compared to healthy controls.

Since LVH develops in a age-dependent manner, genetic diagnosis provides a mechanism for early identification of individuals at risk for developing HCM, prior to the expression of diagnostic clinical manifestations. One goal for the next era of medicine is to evolve from contemporary symptom palliation of late stage disease to early preventive strategies which instead strive to alter the natural history of disease development.

STUDY OBJECTIVES:

The goal of this trial is to evaluate the safety, feasibility, and efficacy of diltiazem administration in attenuating the natural history of HCM, focusing on tolerability and impact on diastolic function. The primary efficacy endpoint will be an improvement in diastolic function in G+/LVH- subjects receiving active therapy as compared to placebo, as measured by improved mean tissue Doppler echocardiographic early diastolic velocity (E') in the diltiazem group compared to the placebo group 2 years after randomization. As a pilot trial, treatment effects on multiple related parameters including changes in LV dimensions and mass, development of overt LVH, development of cardiac magnetic resonance (CMR) evidence of fibrosis, and levels of serum biomarkers will be analyzed in an exploratory manner to more fully characterize potential treatment effect. The safety endpoint will be no excess of all cause death, cardiovascular death (including sudden death), heart failure requiring medication or hospitalization, or a significant difference in the development of symptoms/side effects which necessitate discontinuation of treatment in the active vs placebo arm.

STUDY DESIGN AND SCHEMA A placebo-controlled, randomized double-blind Pilot clinical trial.

Eligible G+/LVH- subjects will undergo baseline studies (physical examination, echocardiography, CMR, blood tests) and will be randomized to receive diltiazem or placebo in a double blind fashion. There is a 3 week titration phase to increase the dose of study drug to target. The total duration of the study protocol is 5 years: study drug will be continued for a total of 4 years and a 1 year post-treatment evaluation will be performed. The primary endpoint will be assessed after 2 years of treatment.

Study visits and data collection consist of echocardiography at 3, 6, 12, 18, 24, 36,48, and 60 months. Annual evaluations consisting of physical exam, echocardiography, EKG, and measurement of serum biomarkers will also be performed.

PATIENT POPULATION Eligible subjects will have an identified sarcomere mutation with no clinical evidence of LVH. Children age 15 years and older will be enrolled at Brigham and Women's Hospital; children age 5-15 years will be enrolled via Children's Hospital Boston.

Major Inclusion Criteria:

* Preclinical HCM as defined by above G+/LVH- criteria
* Able to provide informed consent (or parental consent)

Major Major Exclusion Criteria:

Contraindication to diltiazem administration, including the following pre-existing conditions:

* Second or third degree atrioventricular block
* Symptomatic heart failure
* Sick sinus syndrome
* Concomitant treatment with verapamil and/or beta-blockers
* Concomitant treatment with cyclosporine or FK506
* Impaired hepatic or renal function
* Age <5 years
* Pregnant or breastfeeding women

PRIMARY AND SECONDARY ENDPOINTS

PRIMARY ENDPOINT:

Improvement in diastolic function as reflected by the averaged E' velocity compared to baseline (E' velocities improve, remain stable, or decline less in the treated group) 2 years following initiation of treatment.

As a pilot study, numerous other parameters reflecting myocardial structure and function will also be explored.

SECONDARY ENDPOINTS:

* Development of left ventricular hypertrophy
* Improvement in, stability of, or attenuation of increase in serum biomarkers (e.g., BNP, ST2, PICP, PIIINP, PINP) at 3, 6, and 18 months, annually and at study end
* Improvement in, stability of or attenuation of increase in CMR evidence of myocardial fibrosis

  - Impact on left ventricular morphology, remodeling, and cavity size
* Safety: no excess of all cause death, CV death (including sudden death), heart failure requiring medication or hospitalization; No excess of adverse events
* Tolerability: no excess need to reduce or withdraw study medication; no significant difference in adherence to study medication

ELIGIBILITY:
Inclusion Criteria:

* Preclinical HCM (identified sarcomere mutation with no clinical evidence of left ventricular hypertrophy)
* Able to provide informed consent (or parental consent)

Exclusion Criteria:

* Contraindication to diltiazem administration
* Impaired hepatic or renal function
* Age < 5 years
* Pregnant or breastfeeding women

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y Ho, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Fatkin D, McConnell BK, Mudd JO, Semsarian C, Moskowitz IG, Schoen FJ, Giewat M, Seidman CE, Seidman JG. An abnormal Ca(2+) response in mutant sarcomere protein-mediated familial hypertrophic cardiomyopathy. J Clin Invest. 2000 Dec;106(11):1351-9. doi: 10.1172/JCI11093. PMID 11104788
- [Background] Semsarian C, Ahmad I, Giewat M, Georgakopoulos D, Schmitt JP, McConnell BK, Reiken S, Mende U, Marks AR, Kass DA, Seidman CE, Seidman JG. The L-type calcium channel inhibitor diltiazem prevents cardiomyopathy in a mouse model. J Clin Invest. 2002 Apr;109(8):1013-20. doi: 10.1172/JCI14677. PMID 11956238
- [Background] Ho CY, Sweitzer NK, McDonough B, Maron BJ, Casey SA, Seidman JG, Seidman CE, Solomon SD. Assessment of diastolic function with Doppler tissue imaging to predict genotype in preclinical hypertrophic cardiomyopathy. Circulation. 2002 Jun 25;105(25):2992-7. doi: 10.1161/01.cir.0000019070.70491.6d. PMID 12081993
- [Background] Ho CY, Seidman CE. A contemporary approach to hypertrophic cardiomyopathy. Circulation. 2006 Jun 20;113(24):e858-62. doi: 10.1161/CIRCULATIONAHA.105.591982. No abstract available. PMID 16785342
- [Background] Ho CY, Lakdawala NK, Cirino AL, Lipshultz SE, Sparks E, Abbasi SA, Kwong RY, Antman EM, Semsarian C, Gonzalez A, Lopez B, Diez J, Orav EJ, Colan SD, Seidman CE. Diltiazem treatment for pre-clinical hypertrophic cardiomyopathy sarcomere mutation carriers: a pilot randomized trial to modify disease expression. JACC Heart Fail. 2015 Feb;3(2):180-8. doi: 10.1016/j.jchf.2014.08.003. Epub 2014 Oct 31. PMID 25543971
- [Background] Ho CY, Lopez B, Coelho-Filho OR, Lakdawala NK, Cirino AL, Jarolim P, Kwong R, Gonzalez A, Colan SD, Seidman JG, Diez J, Seidman CE. Myocardial fibrosis as an early manifestation of hypertrophic cardiomyopathy. N Engl J Med. 2010 Aug 5;363(6):552-63. doi: 10.1056/NEJMoa1002659. PMID 20818890
- [Background] Ho CY, Abbasi SA, Neilan TG, Shah RV, Chen Y, Heydari B, Cirino AL, Lakdawala NK, Orav EJ, Gonzalez A, Lopez B, Diez J, Jerosch-Herold M, Kwong RY. T1 measurements identify extracellular volume expansion in hypertrophic cardiomyopathy sarcomere mutation carriers with and without left ventricular hypertrophy. Circ Cardiovasc Imaging. 2013 May 1;6(3):415-22. doi: 10.1161/CIRCIMAGING.112.000333. Epub 2013 Apr 2. PMID 23549607
- [Background] Valente AM, Lakdawala NK, Powell AJ, Evans SP, Cirino AL, Orav EJ, MacRae CA, Colan SD, Ho CY. Comparison of echocardiographic and cardiac magnetic resonance imaging in hypertrophic cardiomyopathy sarcomere mutation carriers without left ventricular hypertrophy. Circ Cardiovasc Genet. 2013 Jun;6(3):230-7. doi: 10.1161/CIRCGENETICS.113.000037. Epub 2013 May 20. PMID 23690394
- [Background] Lakdawala NK, Thune JJ, Maron BJ, Cirino AL, Havndrup O, Bundgaard H, Christiansen M, Carlsen CM, Dorval JF, Kwong RY, Colan SD, Kober LV, Ho CY. Electrocardiographic features of sarcomere mutation carriers with and without clinically overt hypertrophic cardiomyopathy. Am J Cardiol. 2011 Dec 1;108(11):1606-13. doi: 10.1016/j.amjcard.2011.07.019. Epub 2011 Sep 21. PMID 21943931
- [Derived] Ho CY, Cirino AL, Lakdawala NK, Groarke J, Valente AM, Semsarian C, Colan SD, Orav EJ. Evolution of hypertrophic cardiomyopathy in sarcomere mutation carriers. Heart. 2016 Nov 15;102(22):1805-1812. doi: 10.1136/heartjnl-2016-310015. Epub 2016 Sep 2. PMID 27590665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the HCM clinics at Brigham and Women's Hospital (Boston, MA), Boston Children's Hospital (Boston, MA), and Royal Prince Alfred Hospital (Sydney, Australia). Participants were recruited from 2006 through 2010.
Groups:
- I- Diltiazem (Active Arm): Diltiazem: Titrated to a target dose of 360 mg daily (sustained release formulation) for the duration of the study period
Period: Overall Study
Arm/Group | I- Diltiazem (Active Arm) | II- Placebo
Started | 19 | 20
Completed | 18 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled through Brigham and Women's Hospital (Boston, MA), Boston Children's Hospital, and Royal Prince Alfred Hospital (Sydney, Australia) were randomized 1:1 to diltiazem or placebo. Participants were 5-39 years old, carried the sarcomere mutation presumed to cause HCM in the family, and had normal LV wall thickness by echo.
Groups:
- I- Diltiazem: Diltiazem: Titrated to a target dose of 360 mg daily (sustained release formulation) for the duration of the study period
- Total: Total of all reporting groups
Arm/Group | I- Diltiazem | II- Placebo | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.7) | 17.3 (2.1) | 15.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Increase, Stability of, or Decrease in the Decline of Diastolic Function as Reflected by the Global Early Myocardial Relaxation (E') Velocity
Description: The change in E' velocity (difference between final value - baseline value) was compared between participants who received diltiazem and those who received placebo to gauge treatment response. Please note that the total duration on treatment varied between study subjects to maximize time on treatment for the trial. Specifically, subjects that enrolled earliest had the longest duration of treatment; those who enrolled latest had the shortest duration of treatment with a minimum treatment duration of 1 year. All analyses examine the final study visit on treatment to the baseline visit.
Time Frame: Baseline and final study visits
Measure: Mean (Standard Error); unit: cm/sec (difference final-baseline)
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
cm/sec (difference final-baseline) | -0.06 (0.27) | -0.21 (0.42)
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Change in E' Velocity comparing baseline and final study visits; Test type: Superiority or Other; p = 0.75, Generalized estimating equation — Adjusted for age, sex, genotype, family relations, and baseline value. p<0.05 considered statistically significant; Generalized estimating equation approach accounting for an exchangeable correlation structure within families

2. Secondary Outcome: Safety and Tolerability of Diltiazem Treatment
Description: Adverse events were compared between participants assigned to diltiazem and those assigned to placebo
Time Frame: Baseline through final study visits
Measure: Number; unit: Participants Reporting Adverse Events
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
Participants Reporting Adverse Events | 10 | 12
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Adverse Events; Test type: Superiority or Other; p = 0.99, Fisher Exact

3. Secondary Outcome: Impact of Diltiazem on Heart Rate
Description: Change in Value (Difference between Final and Baseline Visits)
Time Frame: Baseline and final study visits
Measure: Mean (Standard Error); unit: beats/minute
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
beats/minute | -4.9 (2.2) | 2.0 (2.6)
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Test type: Superiority or Other; p > 0.06, Generalized Estimating Equation — Adjusted for age, sex, genotype, family relations, and baseline value. p<0.05 considered statistically significant; Generalized estimating equation approach accounting for an exchangeable correlation structure within families

4. Secondary Outcome: Left Ventricular Cavity Size
Description: Change in Left Ventricular End-Diastolic Diameter z-score (Final Value - Baseline Value)
Time Frame: Baseline and final study visits
Measure: Mean (Standard Error); unit: z-score units
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
z-score units | 0.60 (0.17) | -0.53 (0.16)
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Change in LV End-Diastolic Diameter z-score from baseline to final visit; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equation — Adjusted for age, sex, genotype, family relations, and baseline value; Generalized estimating equation approach accounting for an exchangeable correlation structure within families

5. Secondary Outcome: Development of Left Ventricular Hypertrophy
Description: The number of participants who developed overt left ventricular hypertrophy during the duration of the trial was analyzed
Time Frame: Baseline through final study visits
Measure: Number; unit: participants
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
participants | 2 | 2

6. Secondary Outcome: Adherence to Study Medication
Description: Adherence to study medication was assessed by pill count
Time Frame: Duration of the trial
Measure: Median (Standard Deviation); unit: percentage of pills taken
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
percentage of pills taken | 83 (10.8) | 90 (6.6)
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Percentage adherent to study medication; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Impact of Diltiazem on Systolic Blood Pressure
Description: Change in Value (Difference between Final and Baseline Visits)
Time Frame: Baseline and final study visits
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | I- Diltiazem | II- Placebo
Number analyzed (Participants) | 18 | 20
mmHg | -1.4 (1.7) | 2.1 (1.8)
Statistical Analysis 1: Comparison: I- Diltiazem vs II- Placebo; Test type: Superiority or Other; p = 0.15, Generalized estimating equation — Adjusted for age, sex, genotype, family relations, and baseline value; Generalized estimating equation approach accounting for an exchangeable correlation structure within families

ADVERSE EVENTS:
Time Frame: Duration of Trial
Arm/Group | I- Diltiazem | II- Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 10/18 | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I- Diltiazem (N=18) | II- Placebo (N=20)
Shortness of Breath (Cardiac disorders) | 6 (9) | 1 (1)
Lightheadeness (Cardiac disorders) | 3 (5) | 5 (6)
Nausea/GI distress (Gastrointestinal disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Chest Pain (Cardiac disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of participants and short follow-up duration. Currently available tools to monitor treatment response/ phenotypic progression are may lack adequate resolution. The penetrance of sarcomere mutations is variable and may not be complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No